CLINICAL TRIAL: NCT02646189
Title: Therapeutic Safety and Efficacy of REP 2139 (REP 9AC') in HBV Infected Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Replicor Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REP 102
Record Dates: First submitted 2016-01-03; First posted 2016-01-05 (Estimated); Last update posted 2016-01-05 (Estimated); Status verified 2016-01

CONDITIONS: Hepatitis B, Chronic
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — Thymalfasin; peginterferon alfa-2a

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- REP 2139-Ca + immunotherapy (Experimental): REP 2139-Ca is the calcium chelate complex formulation of REP 2139.
  Zadaxin is thymosin alpha 1
  Pegasys is pegylated interferon alpha 2a
  Patients initially receiving REP 2139-Ca with no Grade 3 adverse events at week 20 are eligible to transition to combination therapy with Zadaxin if serum HBV DNA is > 2000 copies / ml.
  After 10 weeks of REP 2139-Ca / Zadaxin combination therapy, patients not experiencing a measurable improvement in serum antiviral response can further transition to combination therapy with REP 2139-Ca and Pegasys.
  Interventions: Drug: REP 2139-Ca; Drug: Zadaxin; Drug: Pegasys

INTERVENTIONS:
Drug: REP 2139-Ca — REP 2139-Ca is administered weekly at 250 or 500mg doses by slow IV infusion.
Drug: Zadaxin — Zadaxin is administered twice weekly (1.6mg) by subcutaneous injection
  Other Names: thymosin alpha 1
Drug: Pegasys — Pegasys in administered once weekly by subcutaneous injection with dose escalation to 180ug / week.
  Other Names: pegylated interferon alpha-2a

SUMMARY:
REP 9AC (REP 2055) is a nucleic acid polymer (NAP) with entry and post-entry antiviral activity against duck hepatitis B virus (DHBV) infection. REP 2055 has been shown to have potent therapeutic effect against established DHBV infection in vivo

REP 2055 was additionally shown to have significant antiviral effects in patients with chronic HBV infection in the previous REP 101 study. REP 2139 is a version of REP 2055 designed for improved administration tolerability and stability.

The safety and antiviral activity REP 2139, first in monotherapy and then in combination with immunotherapy in patients with chronic HBV infection will be assessed in the REP 102 protocol.

DETAILED DESCRIPTION:
Chronic hepatitis B is a long term condition caused by infection of the body with the hepatitis B virus (HBV). This infection often results in inflammation or scarring of the liver and can eventually lead to liver cirrhosis and liver failure. These infections are also one of the major causes of the development of hepatocellular carcinoma (liver cancer).

Although some drugs have been approved to treat chronic hepatitis B infections, they do not provide a complete cure except in rare cases (a cure generally means that a person loses the hepatitis B virus from the blood and the liver and develops a durable immunological control of subsequent HBV infection). However, these drugs do significantly decrease the risk of liver damage and liver cancer arising from the presence of a chronic liver infection by slowing or stopping the production of infectious virus. Thus the primary problem associated with currently available drugs is the lack of clearance of the virus from the hepatocytes which necessitates long term treatment with these drugs. There is clearly a need to identify new drugs that can benefit patients with chronic hepatitis B infections. Nucleic acid-based polymers (NAPs) are a new class of broad-spectrum antiviral compounds which act against HBV infection by blocking the release of the surface antigen protein (HBsAg) from infected hepatocytes. In the human patients in the REP 101 protocol, the previous NAP clinical candidate, REP 9AC (REP 2055), rapidly induced pronounced reductions in or clearance of serum HBsAg in 7 out of 8 patients. HBsAg is the major immunoinhibitory mechanism by which HBV maintains its chronicity and by reducing or eliminating HBsAg from the blood, REP 9AC appears able to elicit restoration of durable immunological responses in patients capable of clearing the HBV infection. The performance of REP 9AC in providing sustained virologic responses (SVRs) in patients with chronic HBV infection appeared to be far superior than any compound currently approved for the treatment of HBV infection

REP 9AC' (REP 2139) is a modified version of its predecessor, REP 9AC (REP 2055). Both are 40mer phosphorothioate oligonucleotides comprised of alternating adenosine and cytidine nucleotides and in the case of REP 9AC, has been shown to have low toxicity and to be highly effective in treating hepatitis B infection in human patients. The modifications in REP 9AC' significantly improve the stability and reduce the pro-inflammatory activity of REP 9AC' compared to that of REP 9AC while retaining all the antiviral activity found in REP 9AC. Both these modifications (5-methylation of cytosines and 2' O methylation of the ribose sugar in each nucleotide) are naturally occurring modifications in human nucleic acid and are known to be well tolerated in clinical trials. It is expected that REP 9AC' will be able to achieve a more robust antiviral activity in patients with chronic HBV with significantly lower dosing requirements and fewer side effects than REP 9AC.

Current interim data analysis from the still ongoing REP 101 assessing the activity of REP 9AC in patients with chronic HBV infection indicates the following:

1. REP 9AC exposure in eight patients has been generally well tolerated at doses up to 600mg / week and 400mg / day (for seven continuous days). Administration related side effects include mild to moderate pro-inflammatory reactions during the drug administration (itching and fever) which disappear after drug administration is complete. Chronic side effects include mild elevations in blood anticoagulation (international normalized ratio ~1.5) and serum hypocalcemia (which is easily mitigated with a mineral supplement).
2. REP 9AC has achieved serum HBsAg reduction or clearance in all patients compliant with the proscribed dosing regimen (7 out of 7).
3. In these seven patients, 5 have demonstrated restoration of at least a partial immunological control of their infection (appearance of serum anti-HBs and the establishment of a lower serum HBV DNA setpoint).
4. Of the five patients achieving having an immunological response, three have achieved a SVR off treatment with as few as 20 weeks of REP 9AC treatment with complete and durable immunological control over their infection for 18, 12 and 10.5 months.
5. Suboptimal stability of REP 9AC is a likely factor impairing the performance of the drug.

This proposed study is designed to demonstrate that REP 9AC' can be well tolerated when given to human patients chronically infected with HBV and to evaluate if a reduction of viral titers can be observed when REP 9AC' is administered as a monotherapy and then in combination with immunotherapy.

NAPs: Replicor's technology utilizes the novel properties of NAPs to inhibit interactions critical for viral activity. This technology is active in vitro against all known families of enveloped viruses. REPLICor's proof of concept compounds, REP 9 (REP 2006) and REP 9C (REP 2031) and its first generation clinical candidate, REP 9AC (REP 2055) have also demonstrated potent antiviral activity in vivo against the following viral infections: HCV, HBV (DHBV), Cytomegalovirus, Herpes Simplex virus-2, Ebola, influenza and respiratory syncytial virus.

NAPs (REP 9, REP 9C and REP 9AC) have been administered at therapeutically active doses in acute and chronic regimens by multiple routes of administration (parenteral, oral, topical and aerosol) in mice, rats, hamsters, guinea pigs, ducks and non human primate species with no detectable side effects. Moreover, this class of chemical compounds (phosphorothioate oligonucleotides) are known to be well tolerated in human patients in several clinical trials.

REPLICor has validated the compatibility of the modifications in REP 9AC' with the antiviral activity present in NAPs indirectly: the 2'O methyl sugar modification was found to not affect the antiviral activity of NAPs against duck hepatitis B virus in vivo and further shown to substantially improve the stability of NAPs to nuclease degradation and substantially reduce their immunoreactivity in human peripheral blood mononuclear cells . The 5'methylation of cytosine was shown not to affect target interaction in cell free interaction assays and is well known to mitigate the immunoreactivity of nucleic acids.

It is now a widely held notion that any successful outcome in the treatment of chronic HBV must involve immunostimulation in order to catalyze restoration of the appropriate immune responses (both adaptive and innate) in order to achieve durable control over HBV infection after therapy. The results from REP 101 protocol suggest that elimination of serum HBsAg removes the chronic immunosuppression mediated by this protein. However there is a heterogeneous immunological response to HBsAg reduction / clearance in the patients treated to date (as measured by serum HBV DNA decline): only about 40% of patients appear to exhibit a strong immunological response after the reduction / removal of serum HBsAg . This observation strongly suggests that while HBsAg suppression is essential for establishing durable immunological control, specific immunostimulation may also be required in many patients in order for them to achieve durable immunological control .

Thymosin alpha 1 (Zadaxin™) is synthetically prepared thymosin alpha 1 polypeptide (28 amino acids, molecular weight 3108) which is identical to the naturally occurring thymosin alpha 1 present in humans. Thymosin alpha 1 shares homology with the interferon alpha family of peptides but unlike interferon alpha, Zadaxin administration in human subjects is not accompanied by any significant side effects. More importantly, Zadaxin administration with other proinflammatory compounds (like interferon alpha) does not alter the side effect profiles of those compounds.

Zadaxin shares many of the immunostimulatory properties of interferon alpha in that it is able to stimulate the production of several cytokines important in reestablishing an immune response capable of controlling the HBV infection. Zadaxin is also able to stimulate the production of natural killer, CD4 and CD8 cells all known to be correlated with the establishment of a durable immunological control of HBV infection.

In the treatment of chronic HBV in the clinic, Zadaxin monotherapy is able to achieve HBeAg and HBV DNA seroclearance in 30-50% of patients which is comparable or better than that achievable with interferon alpha. More important is the consistent observation that the proportion of patients achieving HBV DNA seroclearance off therapy continually increases (an effect not observed with interferon alpha).

Based on the very low side effect profile of Zadaxin (both as a monotherapy and in combination with interferon alpha and HBV polymerase inhibitors) and its clear ability to stimulate functional and durable immune response and control of HBV in patients with chronic HBV infections, the investigators strongly suspect that Zadaxin add-on therapy in patients currently receiving REP 9AC' will be safe and may have a synergistic effect on the ability of patients to achieve durable immunological control, thus greatly increasing the proportion of patients achieving durable immunological control with REP 9AC' - Zadaxin therapy compared to either therapy alone.

It may be possible that the immunostimulation provided by Zadaxin™ may not provide a strong or broad enough immunostimulatory effect to provide an additive or synergistic antiviral response from the patient's immune system while on REP 9AC' therapy. Since Pegasys™ is a much stronger immunostimulatory drug but having significant side effects, dosing with this compound will be slowly escalated each week to a full dose (180 ug once weekly) providing no grade 3 adverse events are observed.

ELIGIBILITY:
Inclusion Criteria:

* HBsAg+
* Anti-HBs negative
* HBV titer > 1x10^7 copies / ml
* Treatment naïve
* HIV / HCV / hepatitis delta virus negative
* Fibrosis with compensation (as determined by Fibroscan and liver enzymes)
* Non cirrhotic
* No known active cytomegalovirus infection
* Willingness to utilize adequate contraception while being treated with REP 9AC' and for 6 months following the end of treatment
* Adequate venous access allowing weekly intravenous therapies and blood tests

Exclusion Criteria:

* Evidence of cardiovascular disease
* Autoimmune hepatitis
* Presence of Wilson's disease
* Presence of severe NAFLD
* Evidence of any other co-existent liver disease
* Anti-nuclear antibody positive
* Evidence of liver cirrhosis
* A history of ascites, hepatic encephalopathy or variceal hemorrhage
* Body weight > 100 kg
* Platelet count < 75,000, polymorphonuclear cell count < 1,500 or hematocrit < 33%
* Alpha feto protein > 100 ng/ml or the presence of a hepatic mass suggestive of hepatocellular carcinoma .
* Bilirubin > 2.5 mg/dl
* Creatinine > 1.5 mg/dl
* Platelet count < 75,000 / cmm
* Serum albumin < 35 mg/ml
* Poorly controlled diabetes mellitus
* Another serious medical disorder
* A serious psychiatric disorder
* Uncontrolled hypertension
* A history of alcohol abuse within the last year
* The use of illicit drugs within the past two years
* Inability to provide informed consent
* Positive pregnancy test
* Breastfeeding
* Inability or unwillingness to provide weekly blood samples
* Poor venous access making IV infusion too difficult

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2011-08; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of REP 2139-Ca + immunotherapy | 40 weeks (treatment)
  To record side effects, symptoms and adverse effects of exposure to REP 2139-Ca in monotherapy and when combined with Zadaxin and / or Pegasys.

SECONDARY OUTCOMES:
Efficacy of REP 2139-Ca + immunotherapy | 40 weeks (treatment) + 52 weeks (follow up)
  To assess antiviral activity of REP 2139-Ca in monotherapy and when combined with Zadaxin and / or Pegasus including serum HBsAg, HBeAg, anti-HBsAg antibodies, anti-HBeAg antibodies and HBV DNA.

CONTACTS AND LOCATIONS:
Overall Officials: Mamun Al-Mahtab, MD, Principal Investigator — Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Locations (1):
- Farabi General Hospital, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Noordeen F, Vaillant A, Jilbert AR. Nucleic acid polymers inhibit duck hepatitis B virus infection in vitro. Antimicrob Agents Chemother. 2013 Nov;57(11):5291-8. doi: 10.1128/AAC.01003-13. Epub 2013 Aug 12. PMID 23939902
- [Background] Noordeen F, Vaillant A, Jilbert AR. Nucleic acid polymers prevent the establishment of duck hepatitis B virus infection in vivo. Antimicrob Agents Chemother. 2013 Nov;57(11):5299-306. doi: 10.1128/AAC.01005-13. Epub 2013 Aug 12. PMID 23939904
- [Background] Noordeen F, Scougall CA, Grosse A, Qiao Q, Ajilian BB, Reaiche-Miller G, Finnie J, Werner M, Broering R, Schlaak JF, Vaillant A, Jilbert AR. Therapeutic Antiviral Effect of the Nucleic Acid Polymer REP 2055 against Persistent Duck Hepatitis B Virus Infection. PLoS One. 2015 Nov 11;10(11):e0140909. doi: 10.1371/journal.pone.0140909. eCollection 2015. PMID 26560490
- [Background] Jiang YF, Ma ZH, Zhao PW, Pan Y, Liu YY, Feng JY, Niu JQ. Effect of thymosin-alpha(1) on T-helper 1 cell and T-helper 2 cell cytokine synthesis in patients with hepatitis B virus e antigen-positive chronic hepatitis B. J Int Med Res. 2010;38(6):2053-62. doi: 10.1177/147323001003800620. PMID 21227010
- [Background] Iino S, Toyota J, Kumada H, Kiyosawa K, Kakumu S, Sata M, Suzuki H, Martins EB. The efficacy and safety of thymosin alpha-1 in Japanese patients with chronic hepatitis B; results from a randomized clinical trial. J Viral Hepat. 2005 May;12(3):300-6. doi: 10.1111/j.1365-2893.2005.00633.x. PMID 15850471
- [Background] Andreone P, Cursaro C, Gramenzi A, Zavagliz C, Rezakovic I, Altomare E, Severini R, Franzone JS, Albano O, Ideo G, Bernardi M, Gasbarrini G. A randomized controlled trial of thymosin-alpha1 versus interferon alfa treatment in patients with hepatitis B e antigen antibody--and hepatitis B virus DNA--positive chronic hepatitis B. Hepatology. 1996 Oct;24(4):774-7. doi: 10.1002/hep.510240404. PMID 8855175
- [Background] Zhuang L, You J, Tang BZ, Ding SY, Yan KH, Peng D, Zhang YM, Zhang L. Preliminary results of Thymosin-a1 versus interferon-alpha-treatment in patients with HBeAg negative and serum HBV DNA positive chronic hepatitis B. World J Gastroenterol. 2001 Jun;7(3):407-10. doi: 10.3748/wjg.v7.i3.407. No abstract available. PMID 11819800
- [Background] You J, Zhuang L, Cheng HY, Yan SM, Yu L, Huang JH, Tang BZ, Huang ML, Ma YL, Chongsuvivatwong V, Sriplung H, Geater A, Qiao YW, Wu RX. Efficacy of thymosin alpha-1 and interferon alpha in treatment of chronic viral hepatitis B: a randomized controlled study. World J Gastroenterol. 2006 Nov 7;12(41):6715-21. doi: 10.3748/wjg.v12.i41.6715. PMID 17075991
- [Derived] Usman Z, Mijocevic H, Karimzadeh H, Daumer M, Al-Mathab M, Bazinet M, Frishman D, Vaillant A, Roggendorf M. Kinetics of hepatitis B surface antigen quasispecies during REP 2139-Ca therapy in HBeAg-positive chronic HBV infection. J Viral Hepat. 2019 Dec;26(12):1454-1464. doi: 10.1111/jvh.13180. Epub 2019 Aug 13. PMID 31323705
- [Derived] Al-Mahtab M, Bazinet M, Vaillant A. Safety and Efficacy of Nucleic Acid Polymers in Monotherapy and Combined with Immunotherapy in Treatment-Naive Bangladeshi Patients with HBeAg+ Chronic Hepatitis B Infection. PLoS One. 2016 Jun 3;11(6):e0156667. doi: 10.1371/journal.pone.0156667. eCollection 2016. PMID 27257978